CLINICAL TRIAL: NCT06024096
Title: Systems Biological Assessment of Statin Effect on Vaccine Responses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Daniel S. Graciaa, MD, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00006239; 2025P010158 (Other: Emory IRB)
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Vaccine Response
Keywords: Flu Vaccine; Statins; Immunization Response; seasonal quadrivalent influenza vaccine; antibody (Ab) response
MeSH Terms: conditions — Influenza, Human | interventions — Atorvastatin; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- seasonal quadrivalent influenza vaccine (QIV) (Active Comparator): Participants will receive the seasonal QIV
  Interventions: Biological: Quadrivalent seasonal influenza vaccine
- statin therapy and a seasonal quadrivalent influenza vaccine (QIV) (Active Comparator): Participants randomized to the Statin + QIV arm will be asked to come back for an extra visit one month prior to the date of vaccination to start statin therapy.
  Interventions: Drug: Atorvastatin; Biological: Quadrivalent seasonal influenza vaccine

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin is a lipid-lowering agent of the statin family that functions by blocking a rate-limiting enzyme, Hydroxymethylglutaryl-CoA (HMG-CoA) reductase, in lipid metabolism. This agent is commonly used for primary and secondary prevention of dyslipidemia. Participants will be asked to take Atorvastatin 80 mg daily at night, for 4 weeks prior to the vaccination, and continue the statin therapy for 4 weeks after vaccination.
  The 80mg dose of atorvastatin allows for evaluation of the immunologic effects of statin medication with a short duration of therapy prior to vaccination.
  Other Names: Statin Therapy
  Arms: statin therapy and a seasonal quadrivalent influenza vaccine (QIV)
Biological: Quadrivalent seasonal influenza vaccine — The FDA-approved quadrivalent seasonal influenza vaccine contains four distinct strains: two influenza A viruses and two influenza B viruses. The approved seasonal QIV will be purchased from the manufacturer to be given for each season of influenza.
  Other Names: Flu vaccine

SUMMARY:
This study is being done to answer the question: Does the use of statin lipid-lowering medication change the effect of influenza vaccine? The research team will use the knowledge gained from answering this question to understand how this medication affects long-lasting immune responses to vaccines. The researchers will study the immune response to the influenza vaccine in the blood (where antibodies are). The team will also look at how statin therapy affects the bacteria that live in the gut by collecting stool samples. To be in this research, participants must be adults willing to receive vaccines.

DETAILED DESCRIPTION:
Statins are widely used for their lipid-lowering and cardiovascular protective effects. Additional research has shown that statins can be anti-inflammatory and play a part in modulating the immune system. These effects are called into action in events such as pneumonia, influenza infection, and sepsis. This study will include a screening visit, a statin therapy initiation visit (if the participant is in the statin therapy group), a vaccination visit, and a series of follow-up visits. The statin medication will be dispensed by the study staff with clear instructions on how to take the medication for two months (one month prior to vaccination, and one month after vaccination). Other study procedures include a collection of medical history and medications taken, a urine pregnancy test for participants who are biologically able to become pregnant, a recording of vital signs, and a collection of any adverse events that the participant experiences during their participation in the study. The stool will be collected in one screening visit, at the vaccination visit, and one follow-up visit. Safety tests to evaluate muscle health and liver function will be obtained as well at screening and for participants selected to receive the statin therapy, at two follow-up visits. Memory Aid will be completed by the participant after vaccination.

The blood and stool samples collected during this study will be stored and tested to evaluate how the immune system responds to statin therapy and vaccination over time. The remaining unused samples will be stored for use in future research.

This research will help advance the knowledge that researchers have on how the immune system reacts to a vaccine if previously exposed to a statin therapy regimen. This will, in turn, enable us to identify the factors that help predict the extent of durability of protection gained from a specific vaccine. This may impact the way future vaccines are developed to provide long-lasting immunity against infections.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and give informed consent.
* Age 18-50 years.
* Women of childbearing potential must agree to use effective birth control for the first 3 months of the study. A negative urine pregnancy test must be documented prior to vaccination.

Exclusion Criteria:

* History of allergy or serious adverse reaction, including Guillain-Barré syndrome, to a vaccine or vaccine products.
* History of a medical condition resulting in impaired immunity such as active solid tumors, leukemia, lymphoma, use of immunosuppressive drugs, chemotherapy, or radiation therapy. Persons with previous skin cancers or cured non-lymphatic tumors are not excluded from the study.
* History of HIV, Hepatitis B, or Hepatitis C infection.
* Chronic clinically significant medical problems that could be considered active or unstable (i.e. diagnosed within the past 3 months or requiring a change in medication within the past 3 months). This includes (but is not limited to):

  1. Insulin-dependent diabetes
  2. Severe heart disease (including arrhythmias)
  3. Severe lung disease
  4. Severe liver disease
  5. Severe kidney disease
  6. Severe hypertension: defined as life-threatening consequences (e.g., malignant hypertension, transient or permanent neurologic deficit).
* BMI > 30
* Current or previous use of statins or any other lipid-lowering drug.
* Pregnancy or breastfeeding or plans to become pregnant in the first 3 months of study participation.
* History of influenza infection within the same influenza season.
* Receipt of blood products or immune globulin products within the prior 3 months.
* History of excessive alcohol consumption, drug use, psychiatric conditions, social conditions, or occupational conditions that in the opinion of the investigator would preclude compliance with the trial.
* Receipt of any live vaccines 30 days before or plans to receive any live vaccines 30 days after vaccination.
* Receipt of any inactivated vaccines 14 days before or plans to receive any inactivated vaccines 14 days after vaccination.

For participants randomized to the statin therapy + QIV group:

* The participant is currently taking any medication that has known interactions with statin therapy.
* History of renal or hepatic impairment.
* Abnormal Safety lab results >1.5 upper limit normal (ULN)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S. Graciaa, MD, MPH, MSc, Principal Investigator — Emory University; Nadine Rouphael, MD, Principal Investigator — Emory University; Varun Phadke, MD, Principal Investigator — Emory University; Vin Tangpricha, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Hope Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will share de-identified participant data (including data dictionaries) and Transcriptomics data.
Supporting Information: Study Protocol
Time Frame: The team will share the data immediately following the study publication.
Access Criteria: Data will be available via NCBI GEO
URL: http://www.ncbi.nlm.nih.gov/geo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Hope Clinic in Atlanta, Georgia, USA. Participant enrollment began September 20, 2023, and all follow-up was completed by December 16, 2024.
Groups:
- Statin Therapy and a Seasonal Quadrivalent Influenza Vaccine (QIV): Participants randomized to the Statin + QIV arm will be asked to come back for an extra visit one month prior to the date of vaccination to start statin therapy.
  Atorvastatin: Atorvastatin is a lipid-lowering agent of the statin family that functions by blocking a rate-limiting enzyme, Hydroxymethylglutaryl-CoA (HMG-CoA) reductase, in lipid metabolism. This agent is commonly used for primary and secondary prevention of dyslipidemia. Participants will be asked to take Atorvastatin 80 mg daily at night, for 4 weeks prior to the vaccination, and continue the statin therapy for 4 weeks after vaccination.
  The 80mg dose of atorvastatin allows for evaluation of the immunologic effects of statin medication with a short duration of therapy prior to vaccination.
  Quadrivalent seasonal influenza vaccine: The FDA-approved quadrivalent seasonal influenza vaccine contains four distinct strains: two influenza A viruses and two influenza B viruses. The approved seasonal QIV will be purchased from the manufacturer to be given for each season of influenza.
Period: Overall Study
Arm/Group | Seasonal Quadrivalent Influenza Vaccine (QIV) | Statin Therapy and a Seasonal Quadrivalent Influenza Vaccine (QIV)
Started | 30 | 33
Completed | 26 | 24
Not Completed | 4 | 9
Not completed — Lost to Follow-up | 2 | 5
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seasonal Quadrivalent Influenza Vaccine (QIV) | Statin Therapy and a Seasonal Quadrivalent Influenza Vaccine (QIV) | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 33 | 63
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.10 (8.10) | 32.67 (7.80) | 32.40 (7.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 12 | 18 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 24 | 32 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 7 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 11 | 20
  White | 15 | 14 | 29
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 33 | 63

OUTCOME MEASURES:

1. Primary Outcome: Magnitude of the Antibody (Ab) Response to QIV in Statin Recipients and Non-recipients.
Description: Magnitude of neutralizing antibody responses against influenza vaccine strains at 29 days after vaccination among participants.
Time Frame: Up to 29 days after vaccine administration
Measure: Geometric Mean (Standard Deviation); unit: log fold-change (logFC)
Arm/Group | Seasonal Quadrivalent Influenza Vaccine (QIV) | Statin Therapy and a Seasonal Quadrivalent Influenza Vaccine (QIV)
Number analyzed (Participants) | 25 | 21
log fold-change (logFC)
  H1N1 | 1.33 (0.36) | 1.46 (0.65)
  H3N2 | 1.35 (0.41) | 1.28 (0.25)

2. Secondary Outcome: Number of Adverse Events (AEs) Grade 2 or Higher
Description: Adverse events of grade 2 or higher (AE, defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of the vaccine, without any judgment about causality) will be identified during questioning or examination of participants during study visits or receiving a safety contact from a participant.
Time Frame: Until day 29 after vaccine administration
Measure: Number; unit: Adverse events
Arm/Group | Seasonal Quadrivalent Influenza Vaccine (QIV) | Statin Therapy and a Seasonal Quadrivalent Influenza Vaccine (QIV)
Number analyzed (Participants) | 30 | 33
Adverse events | 1 | 4

3. Secondary Outcome: Number of Adverse Events (AEs)
Description: Adverse events (AE) will be graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 5.0
Time Frame: Until day 29 after vaccine administration
Measure: Number; unit: Adverse events
Arm/Group | Seasonal Quadrivalent Influenza Vaccine (QIV) | Statin Therapy and a Seasonal Quadrivalent Influenza Vaccine (QIV)
Number analyzed (Participants) | 30 | 33
Adverse events
  Grade 1 | 0 | 0
  Grade 2 | 1 | 3
  Grade 3 | 0 | 1
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAE, defined as an AE that in the view of the investigator results in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect) will be identified during questioning or examination of participants during study visits or receiving a safety contact from a participant any time during the study.
Time Frame: Up to 181 days after vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Seasonal Quadrivalent Influenza Vaccine (QIV) | Statin Therapy and a Seasonal Quadrivalent Influenza Vaccine (QIV)
Number analyzed (Participants) | 30 | 33
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time consent to participate in the study was obtained, through up to 181 days after vaccine administration.
Arm/Group | Seasonal Quadrivalent Influenza Vaccine (QIV) | Statin Therapy and a Seasonal Quadrivalent Influenza Vaccine (QIV)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/33
Other Adverse Events (participants affected / at risk) | 1/30 | 3/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Seasonal Quadrivalent Influenza Vaccine (QIV) (N=30) | Statin Therapy and a Seasonal Quadrivalent Influenza Vaccine (QIV) (N=33)
Vomiting (Grade 2) (Gastrointestinal disorders) | 1 | 0
Elevation in transaminases (Grade 2) (Hepatobiliary disorders) | 0 | 1
Elevation in bilirubin (Grade 2) (Hepatobiliary disorders) | 0 | 1
Elevation in Creatine (Grade 2) (Renal and urinary disorders) | 0 | 1
Elevation in Creatine Kinase (Grade 3, asymptomatic) (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT06024096/Prot_SAP_000.pdf